CLINICAL TRIAL: NCT04738227
Title: Effect of Low-level Laser Therapy on Salivary Flow, pH and Quality of Life in Irradiated Oropharyngeal Cancer Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ziauddin University (Other)
Responsible Party: Principal Investigator, Dr. Danial Arshad, Principal Investigator, Ziauddin University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2480820DAOM
Record Dates: First submitted 2021-02-01; First posted 2021-02-04 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Xerostomia
MeSH Terms: conditions — Xerostomia | interventions — Low-Level Light Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Low level Laser Therapy Group (Experimental): Laser therapy will be performed with a continuous wave diode laser device previously calibrated by the manufacturer.
  6 points that will be the skin overlying the right hand side parotid gland and 3 points on the skin overlying the location of the right hand side submandibular gland).
  Following are the parameters which will be employed for the laser:
  Wavelength - 635nm (visible spectrum), Output power 100 milliwatt, Mean dose per point - 3 J/cm2 , Irradiation time per point 15 s Energy per point 3 J Energy per session 60 J , Laser spot tip will be 0.08cm2 Two laser sessions will be done each week, during 12 weeks, which will bring the total number of laser sessions to All the major salivary glands will be treated with the tip of the laser hand-piece in contact with patients tissues.
  A sum total of 22 points will receive LLLT per session involving all three major salivary glands.
  Interventions: Radiation: Low-Level Laser Therapy

INTERVENTIONS:
Radiation: Low-Level Laser Therapy — Low level laser will be applied and post laser results will be seen to assess any improvements.

SUMMARY:
There are multiple treatment modalities for head and neck cancer. They include radiation therapy, chemotherapy and surgery. Radiation therapy aims to control the tumor with minimum damage to adjacent tissues. Surgery is the preferred treatment for accessible cancers. Radiation and/or chemotherapy is used as an adjunct to surgery, in inaccessible tumors, post surgery sterilization and palliation.

A major complication of RT is that adjacent normal tissues are variably affected.

For Oropharyngeal cancer, major and minor salivary glands are damaged by RT since they fall in the radiation pathway. Atrophy and acinar degeneration are features most commonly found histologically.

Xerostomia is defined as dry mouth resulting from reduced or absent saliva flow.

Xerostomia is not a disease, but may be a symptom of various medical conditions, a side effect of a wide variety of medications and a side effect of a radiation to the head and neck.The flow rate of normal unstimulated saliva is 0.3-0.5 ml/min. If it decreases to less than 0.1-0.2 ml/min, one would experience xerostomia.

According to researchers, the decrease in saliva and xerostomia that results from radiotherapy plays an important role in worsening Quality of Life(QoL) among patients who undergo radiotherapy for head and neck cancers.

Low level laser Therapy(LLLT) uses light energy in the form of photons to produce cellular responses in the cell. Light photons are absorbed by cytochromes and porphyrins in the mitochondria of the cell.

This study aims to prove that Low level laser therapy will improve salivary flow rate, pH and the quality of life in patients who have undergone Radiation therapy for oropharyngeal cancers.

DETAILED DESCRIPTION:
There are multiple treatment modalities the cancers of the head and neck. The main three major treatment options are surgery, radiation therapy and chemotherapy. Radiation therapy (RT) is used to control the growth of the tumor with limiting the damage to adjacent tissues. Surgery is the main treatment for oropharyngeal cancers, but if the cancer remains, radiation and chemotherapy is used in adjunct to surgery. Radiation therapy is a common treatment options for initial to mid stage malignancies.

A major complication of RT is that non neoplastic tissues of the head and neck are variably affected. The exact amount of damage to healthy tissues depends on factors such as fraction of radiation dose, the total amount of the radiation dose administered, volume of irradiated tissue, and how the dose is distributed in the tissue. The effect on the tissues may appear either during the treatment (acute) or once the treatment is complete (late).

For Oropharyngeal cancer, major and minor salivary glands are mostly affected by RT due to the fact that salivary glands fall in the radiation pathway. The mechanisms by which the tissues and cells are damaged due to radiation are still not very clear, but the features most commonly found histologically are atrophy of the tissues and degeneration of the acini. According to researchers, "the decrease in saliva and xerostomia that results from radiotherapy plays an important role in worsening Quality of Life (QoL) among patients who undergo radiotherapy for head and neck cancers". The normal flow rate of unstimulated saliva is 0.3-0.5 ml/min. If it decreases to less than 0.1-0.2 ml/min, it is then that one would experience xerostomia Xerostomia Inventory (XI) which was formulated by Thomson is a validated tool which will also be used to determine the amount of dryness based on the XI score. A higher score will be suggestive of worsening xerostomia.

The most commonly recommended treatment for xerostomia currently is intraoral topical agents. These include salivary stimulants, chewing gums, topical sprays containing malic acid. Also used for xerostomia are medicines such has pilocarpine and cevimeline but both medicines are parasympathomimetic and need to be administered with extreme caution. The effectiveness of there medicines is short lived and only provide symptomatic relief.

Generally, the mechanism by which Low level laser Therapy(LLLT) works is that photons are generated through the light energy and these photons produce cellular responses in the cell. The photons of light are readily absorbed by the cytochromes and the porphyrins present in the mitochondria of the cell.

Low level laser therapy has many diverse effects on the tissues and cells of the body. Previous experimental animal studies highlight a positive effect on the salivary glands when low level laser therapy was applied. Mitotic activity was seen to be stimulated by LLLT to quite an extent in the epithelial tissue of salivary glands of murine test subjects. As a result, the salivary flow rate (SFR) increased, the enzymatic activity increased in saliva significantly as there was a decrease in the activity of peroxidase and catalase enzymes and it was shown to alter the protein concentration in saliva [14,15]. Once the cells receive the LLLT, are more acidic because of the lowered redox state, but soon after the laser therapy they become alkaline resulting in optimal function. Healthy cells are not affected by LLLT as it does not increase their redox potential.

One of the most common side effect of radiation therapy for the oropharyngeal region is Xerostomia. Xerostomia leads to a significant decrease in oral health causing mucositis, dental caries, oral ulcers, periodontal infections etc. These symptoms result in a decrease in the QoL of the patients treated with radiation therapy for oropharyngeal cancers. The conventional treatment for xerostomia is short term symptomatic relief. There is an utmost need for long term treatment that saves the patients from relying on short term treatments.

Objective To determine the effect of low level laser therapy on saliva flow rate in patients who have undergone Radiation therapy for oropharyngeal cancers.

To determine the effect of low level laser therapy on pH of saliva produced in patients who have undergone Radiation therapy for oropharyngeal cancers.

To determine the effect of low level laser therapy on Quality of Life (QoL) in patients who have undergone Radiation therapy for oropharyngeal cancers.

Rationale of the Study Previous studies used a higher wavelength diode laser (808 and 980nm) with controversial results. Some showed excellent results whereas some showed no results at all. The rationale behind choosing a lower wavelength (635nm) in our study is the potentially higher beneficial absorption, to functionally stimulate the damaged, residual salivary glands. No study has been conducted on this particular topic in the Indo-Pak region. Hence, effects of LLLT on salivary glands need to be evaluated.

Significance of the Study As head and neck cancers are increasing in Pakistan, the role of radiation therapy has increased. The side effects of radiation to healthy tissues such as the salivary glands causes severe impairment of oral health and overall quality of life. Low level laser therapy is a relatively non-invasive, cost effective and a new method for treating patients with xerostomia due to radiation therapy. By stimulating residual salivary tissue it may provide long term or permanent (as against symptomatic) relief.

The research would be will be conducted in Karachi, Pakistan where all the facilities of the Laser are available. The procedure will also be done under the supervision of my clinical supervisor, who is a Laser Safety Officer authorized to conduct laser procedures. The patients will be recruited from Ziauddin Hospital where the patients were successfully treated with radiotherapy for oropharyngeal cancers.

Target population The target population will be patients treated with radiotherapy for oropharyngeal cancer in Karachi, Pakistan

Duration of study The duration of study will be 1 year from the date of approval from the Board of advanced studies and research.

The experimental time period will be 12 weeks in which the Patients will be given LLLT two times a week. Each patient would be called at 9am in the morning each day and each patient will have their schedule through out the week so overlapping can be minimized.

Procedure Laser therapy will be performed with a continuous wave diode laser device previously calibrated by the manufacturer.

6 points that will be the skin overlying the right hand side parotid gland and 3 points on the skin overlying the location of the right hand side submandibular gland).

Following are the parameters which will be employed for the laser:

Wavelength - 635nm (visible spectrum), Output power 100 milliwatt, Mean dose per point - 18.75 J/cm2 , Irradiation time per point 15 s Energy per point 3 J Energy per session 33 J , Laser spot tip will be 0.08cm2 Two laser sessions will be done each week, during 12 weeks, which will bring the total number of laser sessions to All the major salivary glands will be treated with the tip of the laser hand-piece in contact with patients tissues.

A sum total of 22 points will receive LLLT per session involving all three major salivary glands.

Parameters to be assessed Three parameters will be assessed

1. Stimulated and Unstimulated salivary flow
2. pH
3. Quality of Life using University of Washington Quality of Life questionnaire

ELIGIBILITY:
Inclusion Criteria:

* Patients with radiation induced persistent xerostomia which will be confirmed clinically and by taking salivary flow rate. Patients which will have salivary flow rate less than 0.1-0.2 ml/min shall be included.
* Patients treated with therapeutic RT for oropharyngeal cancers 3 to 36 months ago
* Patients whose age was equal to or more than 18 years irrespective of gender.

Exclusion Criteria:

* Patients with other determined causes of xerostomia which have been confirmed. Systemic conditions (specially checking and excluding patients having dehydration,patients with known diseases of salivary glands, salivary glands removal surgery, smoking, diabetes, and autoimmune disorders among such as Sjögren's syndrome and drugs that cause xerostomia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2020-11-06 (Actual); Primary Completion 2021-02-03 (Actual); Study Completion 2021-02-03 (Actual)

PRIMARY OUTCOMES:
Increase in Salivary flow rate | 12 weeks
  Increase in salivary flow rate in patients who have undergone Radiation therapy for oropharyngeal cancers.
Increase in pH | 12 weeks
  Increase in pH in patients who have undergone Radiation therapy for oropharyngeal cancers.
Increase in Quality of Life questionnaire Score | 12 weeks
  Increase in the quality of life in patients who have undergone Radiation therapy for oropharyngeal cancers.
  The questionnaire has 13 close ended questions. The total score of the questionnaire will be between 0-1300 A higher score will indicate improvement in the quality of life and will be compared with the score taken at baseline, before the start of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Danial Arshad, M.Phil, Principal Investigator — Ziauddin University
Locations (1):
- Ziauddin University, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No